CLINICAL TRIAL: NCT01762865
Title: Acute Bronchitis in Korea:Associated Microorganisms and Clnincal Findings.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: KOREAABS
Record Dates: First submitted 2013-01-06; First posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Acute Bronchitis
Keywords: acute bronchitis, bacteria, virus, clinical symoptoms
MeSH Terms: conditions — Bronchitis; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum specimens for microbiologic tests

SUMMARY:
The investigators hypothesized that acute bronchitis will be associated with various bacteria and viruses.

DETAILED DESCRIPTION:
The investigators will investigate various bacteria and viruses from colleced specimens from patients with acute bronchitis, and also investigate an assoication of the miroorganims with clinical findings

ELIGIBILITY:
Inclusion Criteria:

* Adults patients aged over 18 years.
* Patients who complain of recent sputum and cough.

Exclusion Criteria:

* Patinets who took antibiotics within 7 days.
* Patinets whose symptoms last for < 5 days.
* Patients who have definite cause of acute cough such as pneumonia, allergic rhinnits, sinusitis, GERD and drug.
* Immunocompromised patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patinets who visit hospitals for recent sputum and/or cough
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Microorganisms (bacteria and/or viruses) related to acute bronchitis | Outcome measure is just type of microoganisms from collected specimens at hospital visit

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Suck Jung, MD, PhD, Principal Investigator — Pulmonary, Allgery and Critical Care Medicine; Hallym University Sacred Heart Hospital
Locations (3):
- South Korea (3):
  - Chunchon Sacred Heart Hospital, Chunchon, Gangwon-do
  - Pumonary, Allegry and Critical Care Medicine; Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Kandong Sacred Heart Hospital, Seoul, Seoul